CLINICAL TRIAL: NCT01531829
Title: Low Dose Rt-PA Plus LMWH Compared With LMWH Alone for the Treatment of Normotensive Pulmonary Embolism Patients With Acute RV Dysfunction: A Randomized，Multi-Center，Controlled Trial
Brief Title: Low Dose Rt-PA for Acute Normotensive Pulmonary Embolism With RVD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Chen WANG, Professor of respiratory and critical care medicine, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJCYH1893
Record Dates: First submitted 2012-02-09; First posted 2012-02-13 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Pulmonary Thromboembolisms; Pulmonary Embolism
Keywords: pulmonary embolism; right ventricular dysfunction; Thrombolysis; Heparin
MeSH Terms: conditions — Pulmonary Embolism; Ventricular Dysfunction, Right | interventions — Tissue Plasminogen Activator; Heparin, Low-Molecular-Weight; Nadroparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose (50mg/2h) rt-PA plus LMWH (Experimental): Low dose (50mg/2h) recombinant tissue plasminogen activator (rt-PA) plus low molecular weight heparin(LMWH)regimen
  Interventions: Drug: Recombinant tissue plasminogen activator (rt-PA)
- LMWH (Active Comparator): Low molecular weight heparin
  Interventions: Drug: Low Molecular Weight Heparin

INTERVENTIONS:
Drug: Recombinant tissue plasminogen activator (rt-PA) — Low dose (50mg/2h) rt-PA plus LMWH
  Other Names: rt-PA
  Arms: Low dose (50mg/2h) rt-PA plus LMWH
Drug: Low Molecular Weight Heparin — 0.1ml/10kg,q12h,5-7 days
  Other Names: Nadroparin
  Arms: LMWH

SUMMARY:
In selected patients with acute pulmonary embolism(PE), low dose (50mg/2h) recombinant tissue plasminogen activator (rt-PA) regimen had been reported to have less bleeding tendency than the FDA-approved rt-PA 100mg/2h regimen 100mg/2h regimen (3% vs.10%), it is worthwhile to reveal whether low dose rt-PA plus low molecular weight heparin (LMWH) can rapidly reverses RV pressure overload in PE, but not increase bleeding and other adverse events. The aim of the study is to compare thrombolytic treatment with LMWH in patients with acute normotensive PE with right ventricular dysfunction(RVD).

DETAILED DESCRIPTION:
In acute pulmonary embolism (PE), normotensive patients with acute RV dysfunction on echocardiography or computed tomography and with myocardial troponin elevation may have an adverse outcome. Thrombolysis rapidly reverses RV pressure overload in PE, but it increases the possibility of bleeding and it remains unclear whether it may improve the early or long-term clinical outcome of these selected normotensive patients.

In our previous study, we found that low dose (50mg/2h) recombinant tissue plasminogen activator (rt-PA) regimen had less bleeding tendency than the 100mg/2h regimen (3% vs.10%), it is worthwhile to reveal whether low dose rt-PA plus Low Molecular Weight Heparin (LMWH) can rapidly reverses RV pressure overload in PE, but not increase bleeding and other adverse events.

In this prospective, multicenter, randomized, control study, we compare low dose rt-PA plus LMWH vs. LMWH alone in acute normotensive pulmonary embolism patients with RV dysfunction. The primary efficacy outcome is the composite of death from any cause or treatment failure, improvements of right ventricular functions on echocardiogram and pulmonary artery obstruction on CT angiographs within 7 days of randomization. Second efficacy outcome is the recurrence of pulmonary embolism and deep venous thrombosis. Safety outcomes include serious life threatening bleeding such as cerebral hemorrhage and other major bleeding episodes, also include mild bleeding. In addition, 90-day clinical and echocardiographic follow-up will be performed, the recurrence of pulmonary embolism and deep venous thrombosis will be recorded. The study is expected to enroll approximately 460 patients.

By determining the benefits vs risks of Low dose rt-PA plus LMWH compared with LMWH alone for the treatment in submassive or intermediate-risk PE, this trial is expected to reveal the worth of Low dose rt-PA plus LMWH treatment and what kind of PE patients are suitable for thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

1. 18 y≤Age≤75y
2. Acute PE (first symptoms occurred 14 d or less before randomization) confirmed by lung scan, or a positive computed tomographic pulmonary angiogram, or a positive selective pulmonary angiogram
3. Hemodynamic stability, diastolic pressure>90mmHg.
4. RV dysfunction confirmed by echocardiography (≥1 criterion), except left-side heart disease, congenital heart disease and mitral valve disease.

   * Increase of the right ventricle showed presented with RV end-diastolic anteroposterior diameter >25 mm, Right/left ventricular end-diastolic diameter >1 (apical or subcostal 4-chamber view) or Right/left ventricular end-diastolic anteroposterior diameter >0.5
   * Hypokinesis of RV-free wall (range of motion less than 5 mm)
   * Tricuspid regurgitation pressure >30mmHg

Exclusion Criteria:

1. RV anterior wall thickness > 5mm confirmed by echocardiography
2. Active internal bleeding and spontaneous intracranial hemorrhage in preceding 6 months
3. Major surgery, organ biopsy or non-compressible punctures within 2 weeks
4. Ischemic stroke occurred within 2 months
5. Gastrointestinal bleeding within 10 days
6. Severe trauma occurred within15 days
7. Neurosurgery or eye surgery within 1 months
8. Severe hypertension difficult to control (systolic blood pressure>180mmHg or diastolic blood pressure>110mmHg)
9. Cardiopulmonary resuscitation
10. Platelet count less than 100×109 / L
11. Pregnancy, or within 2 week post partum
12. Infective endocarditis; left atrial thrombus; aneurysm
13. Serious liver and kidney dysfunction
14. Diabetic hemorrhagic retinopathy
15. Suffering with bleeding disorders
16. Chronic thromboembolic pulmonary hypertension
17. Moderate to severe chronic obstructive pulmonary disease (COPD).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
the composite end point of death from any cause or treatment failure,recurrence of VTE | 7 days
improvements of right ventricular functions on echocardiogram and pulmonary artery obstruction on CT angiographs | 7 days
serious life threatening bleeding such as cerebral hemorrhage and other major bleeding episodes | 7 days
clinical relevant non-major bleedings | 7 days

SECONDARY OUTCOMES:
the composite end point of death from any cause or treatment failure,recurrence of VTE | 3 months and 6 months
improvements of right ventricular functions on echocardiogram and pulmonary artery obstruction on CT angiographs | 3 months and 6 months
serious life threatening bleeding such as cerebral hemorrhage and other major bleeding episodes | 3 months and 6 months
clinical relevant non-major bleedings | 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, PhD,MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (35):
- China (35):
  - Beijing Chao Yang Hospial, Beijing, Beijing Municipality
  - Beijing Daxing People's Hospital, Beijing, Beijing Municipality
  - Beijing Fuwai Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Ministry of Health, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhongshan University in Guangzhou, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Zhongshan University in Guangzhou, Guangzhou, Guangdong
  - The Guangxi Zhuang Autonomous Region people's Hospital, Nanning, Guangxi
  - Guangzhou Shenzhen People's Hospital, Shenzhen, Guangzhou
  - Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - The first hospital of Handan city Hebei Province, Handan, Hebei
  - Hebei Hengshui international Heping Hospital, Hengshui, Hebei
  - Hebei Affiliated Hospital of North China Coal Medical University, Shijiazhuang, Hebei
  - Hebei Medical University Second Hospital, Shijiazhuang, Hebei
  - No.2 Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Third Affiliated Hospital of Inner Mongolia Medical College, Baotou, Inner Mongolia
  - Hospital of Inner Mongolia Autonomous Region, Hohhot, Inner Mongolia
  - Anshan Iron and Steel Company General Hospital, Anshan, Liaoning
  - The first hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - Shenyang Medical College affiliated Fengtian Hospital, Shenyang, Liaoning
  - Affiliated Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The Fourth Military Medical University, Xijing Hospital, Xi'an, Shan'xi
  - Shandong Jining Medical University Affiliated Hospital, Jining, Shandong
  - Shandong Medical College Affiliated Hospital of Qiingdao University, Qingdao, Shandong
  - Shandong Yantai city Yantai Mountain hospital, Yantai, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Second Military Medical University Changhai Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Shanghai Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Medical University Second Hospital, Taiyuan, Shanxi
  - The first hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Sichuan University, West China Hospital, Chengdu, Sichuan
  - The first hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Xinjiang Uygur Autonomous Region people's Hospital, Ürümqi, Xinjiang
  - Zhejiang Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical College in Zhejiang, Wenzhou, Zhejiang